CLINICAL TRIAL: NCT00452660
Title: A Phase IV , Multicenter ,Open Label ,Non Comparative ,Investigator Initiated Study , Evaluating the Effect of Exjade on Oxidative Stress in Low Risk Myelodysplastic Syndrome Patients With Iron Over Load
Brief Title: Evaluation the Effect of Exjade on Oxidative Stress in Low Risk Myelodysplastic Syndrome Patients With Iron Over Load
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other); Tel-Aviv Sourasky Medical Center (Other Government); Sheba Medical Center (Other Government); Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, eliezer rachmilewitz, Head of Hematology Department , E. Wolfson Medical center ,Holon- Israel., Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2412-HMO-CTIL
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: IRON; oxidative stress; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- evaluating the effect of -Exjade (Experimental): evaluating the effect of -Exjade (Deferasirox)_on oxidative stress parameters of blood cells in patients with Low risk Mylodysplastic syndrome ( MDS) with Iron over load
  Interventions: Drug: Exjade

INTERVENTIONS:
Drug: Exjade

SUMMARY:
Certain percentage of MDS patients develop iron overload. Iron is known to participate in intracellular reactions that generate free radicals, inducing oxidative stress and apoptosis, which was found to be increased in MDS patients and consequently resulted in ineffective hematopoiesis. The aim of this study is to evaluate the antioxidant effect of the oral iron chelator Deferasirox -Exjade in low risk MDS patients with iron over load by evaluating changes in several oxidative stress parameters Certain percentage of MDS patients develop iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myelodysplastic syndrome with an IPSS score being Intermediate-1 or low.
* Patients who already received ≥20 unit (100 mL/kg) of packed red blood cells and showing evidence of iron overload (serum ferritin >1000 µg/L).
* Patients post stem cells transplantation with disease recurrence with MDS IPSS score low or intermediate 1.
* Patients who have given consent personally in writing

Exclusion Criteria:

* Patients with myelodysplastic syndrome with an IPSS score being Intermediate-2 or High.
* Patients with serum creatinine >2.0 x ULN
* Patients with ALT(SGPT) levels > 5 x ULN
* Significant proteinuria as indicated by a urinary protein/creatinine ratio >0.5 mg/mg in a non-first void urine sample on two assessments during the screening period.
* History of HIV positive test result. When there are any signs or symptoms indicative of the disease even if the diagnosis is not made, additional test should be conducted.
* History of clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive and ALT above the normal range)
* Patients with systemic uncontrolled hypertension
* Patients with unstable cardiac disease not controlled by standard medical therapy
* Systemic disease (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy or breast feeding. Female of child-bearing potential should conduct contraception during the clinical trial.
* Patients treated with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* Patients being considered by the investigator potentially unreliable and/or not cooperative with regard to the study protocol
* History of hypersensitivity to any of the study drug or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the antioxidative effect of Exjade therapy in MDS patients | one year
with iron over load by evaluating oxidative stress parameters | one year
pre and post treatment | one year

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Exjade over the treatment period. | one year
To analyze iron overload after Exjade treatment period. | one year
To evaluate transfusion requirements. | one year
To confirm the value of LPI, LIP, and Hepcidin as a marker for accurate monitoring of chelation therapy in MDS patients with iron over load. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rachmilewitz Eliezer, MD, Study Chair — Wolfson Medical Center
Locations (1):
- Wolfsom Medical Center, Holon, Israel

REFERENCES:
- [Derived] Ghoti H, Fibach E, Merkel D, Perez-Avraham G, Grisariu S, Rachmilewitz EA. Changes in parameters of oxidative stress and free iron biomarkers during treatment with deferasirox in iron-overloaded patients with myelodysplastic syndromes. Haematologica. 2010 Aug;95(8):1433-4. doi: 10.3324/haematol.2010.024992. Epub 2010 Apr 26. No abstract available. PMID 20421274